CLINICAL TRIAL: NCT03073278
Title: Phase I Feasibility Trial of Stereotactic Re-irradiation of Prostate Cancer Recurrence Within the Definitively Irradiated Prostate
Brief Title: Focal Radiotherapy for Previously Treated Prostate Cancer Patients
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Royal North Shore Hospital (Other)
Collaborators: Northern Sydney and Central Coast Area Health Service (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: Focal SBRT prostate
Record Dates: First submitted 2017-02-27; First posted 2017-03-08 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2026-02

CONDITIONS: Locally Recurrent Prostate Cancer
MeSH Terms: interventions — Radiosurgery

STUDY DESIGN:
Intervention Model Description: Group 1 will receive 36 grays (radiation dose unit Gy) in 6 treatments. Group 2 will receive 38 grays (Gy) in 6 treatments and Group 3 will receive 40 grays (Gy) in 6 treatments. If the first group of participants tolerate the treatment well and with minimal side effects, then the next group of participants will be given the same treatment but at the higher dose (38 Gy). If the second group tolerates this higher dose, then the third group of patients will be given a higher dose (40 Gy). This will be the final dose being tested in this investigation.
Masking Description: no masking
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group 1 (Other): This group of 12 patients will be given 36Gy of Stereotactic Body Radiotherapy (SBRT) divided into six separate doses. This will be delivered two to three time per week.
  Interventions: Radiation: Stereotactic Body Radiotherapy
- Group 2 (Other): This group (12 patients) will be given 38Gy of Stereotactic Body Radiotherapy (SBRT) divided into six separate doses. This will be delivered two to three time per week.
  Interventions: Radiation: Stereotactic Body Radiotherapy
- group 3 (Other): This group (12 patients) will be given 40Gy of Stereotactic Body Radiotherapy (SBRT) divided into six separate doses. This will be delivered two to three time per week.
  Interventions: Radiation: Stereotactic Body Radiotherapy

INTERVENTIONS:
Radiation: Stereotactic Body Radiotherapy — Each group will have different dose of stereotactic body radiotherapy (SBRT). Depending on which group patients are in.

SUMMARY:
To examine the feasibility, safety and toxicity of focal stereotactic radiation treatment (SBRT) for locally recurrent prostate cancer.

DETAILED DESCRIPTION:
Participants must have biopsy proven locally recurrent prostate cancer. Biopsy will be performed by a Urologist. Participants will have PSMA-PET (prostate-specific membrane antigen and positron emission tomography) scan and MRI in Radiology and Nuclear Medicine by experienced Radiologists in the Royal North Shore Hospital. before starting stereotactic radiotherapy. Participants will require fiducial markers inserted in the prostate and may require hydrogel insertion depending on the location of the recurrence. If these are required, it will be done by experienced radiation oncologists. Fiducial markers insertion involves inserting three gold markers into the prostate. It will be used to locate the prostate accurately during radiation treatment. Hydrogel is a temporary gel being injected into the space between the prostate and rectum to reduce the dose of radiation received by the rectum to minimise side effects from the treatment, Focal Stereotactic Body treatment (SBRT) will be used in the study. There are three groups of participants. Each group will receive different level of radiation dose to test the safety of increasing radiation dose. Group 1 will receive 36 grays (radiation dose unit, Gy)) in 6 treatments. Group 2 will receive 38 grays in 6 treatments and Group 3 will receive 40 grays in 6 treatments. The incremental dose escalation will cease if any excess acute toxicity or late grade 3 toxicity. SBRT will be delivered two to three times per week, every second day. The number of treatments per week will depend on the day of the week participants start their treatment. Participants will be reviewed weekly or second weekly. Toxicity will be recorded. A Safety Committee will be formed containing multi-disciplinary team members. All serious adverse events will be reported to the Principal Investigator and Human Research Ethics Committee within 24 hours.

ELIGIBILITY:
Inclusion Criteria:

* Men > 4yrs from external beam radiotherapy (EBRT) meeting the Phoenix definition of biochemical failure or men > 5yrs from EBRT if neo-adjuvant and/or adjuvant androgen deprivation therapy (ADT) also used
* Recurrence localised to less than 1 lobe of prostate on both PMSA and multi-parametric MRI (less than equal to cT2a)
* Recurrence must be biopsy proven, with positive biopsies limited to the PET and MRI suspicious region.
* Life expectancy at least 10yrs from time of SBRT
* PSA < 10

Exclusion Criteria:

* Recurrence in immediate proximity to rectum (unless able to have hydrogel)
* Grade 3 or more toxicity from previous EBRT
* Contra-indicated for fiducial insertion
* GS 8,9 or 10 disease previously (relative - consider if decent disease free interval)

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2017-04-24 (Actual); Primary Completion 2027-03-31 (Estimated); Study Completion 2027-03-31 (Estimated)

PRIMARY OUTCOMES:
feasibility of SBRT dose escalation. This will be assessed by the number of participants with grade 3 acute toxicity according to CTCAE version 4.3 | at weekly review through completion of each radiothrapy dose level, approximately one year
  acute toxicity will be assessed weekly during treatment period to check whether dose escalation can be achieved
safety of SBRT dose escalation. This will be assessed by the number of participants with grade 3 acute toxicity according to CTCAE version 4.3 | at weekly review through completion of each radiothrapy dose level, approximately one year
  outcome will be assessed by reviewing toxicity weekly during the treatment period and at the end of each dose escalation
Toxicity. This will be assessed by the number of participants with grade 3 acute toxicity according to CTCAE version 4.3 and RTOG toxicity score. | at weekly review through completion of each radiothrapy dose level, approximately one year
  outcome will be assessed by reviewing toxicity weekly and at the end of each dose escalation

SECONDARY OUTCOMES:
Tolerability of conservation dose escalation in this cohort of patients | After each group of patients have completed radiotherapy and at 12 and 24 months follow-up. Patients will have routine follow-up 6 monthly for 1 year and then yearly for 10 years post treatment. But study outcomes will only be collected for 2 years.
  outcome will be assessed by reviewing toxicity weekly or secondly weekly and at the end of each dose escalation

CONTACTS AND LOCATIONS:
Overall Officials: George Hruby, Principal Investigator — Northern Sydney Local Health District
Locations (1):
- Royal North Shore Hospital, St Leonards, New South Wales, Australia

IPD SHARING:
Plan to Share IPD: Yes
aim to present data in conferences and publications